CLINICAL TRIAL: NCT06739122
Title: A Phase 3, Open-Label, Multicenter, Single-Arm Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Dulaglutide 3.0 mg and 4.5 mg in Pediatric Participants 10 to Less Than 18 Years of Age With Type 2 Diabetes Mellitus
Brief Title: A Study of Dulaglutide (LY2189265) 3.0 mg and 4.5 mg in Pediatric Participants With Type 2 Diabetes Mellitus (AWARD-PEDS PLUS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27198; H9X-MC-GBGS (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dulaglutide (Experimental): Participants will receive dulaglutide subcutaneously (SC)
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265

SUMMARY:
The main purpose of this study is to evaluate additional dosing options for dulaglutide in pediatric participants with Type 2 Diabetes. Participation in this study will last about 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 diabetes treated with diet and exercise and metformin and/or basal insulin. Metformin and/or basal insulin dose must be stable for at least 8 weeks prior to screening.
* Have a body weight ≥50 kilograms (kg) and Body Mass Index (BMI) of >85th percentile

Exclusion Criteria:

* Have Type 1 diabetes
* Have received treatment with any glucose-lowering agent(s) other than metformin or basal insulin within 8 weeks prior to screening
* After the Type 2 diabetes diagnosis, have a history of diabetic ketoacidosis or hyperosmolar syndrome
* Have had ≥1 episode of severe hypoglycemia and/or ≥1 episode of hypoglycemic unawareness within the last 6 months
* Have family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2)
* Have prior chronic, recurrent, or idiopathic pancreatitis, or known gallbladder disease
* Have been treated with prescription drugs or over-the-counter medications that promote weight loss within 8 weeks prior to screening

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Events (SAE) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 26
  A summary of treatment emergent adverse events (TEAEs), SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Dulaglutide | Predose through Week 30
PK: Maximum Observed Concentration (Cmax) of Dulaglutide | Predose through Week 30
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 26
Percent Change from Baseline in Body Weight | Baseline, Week 26
Change from Baseline in Total Cholesterol | Baseline, Week 26
Change from Baseline in the EQ-5D-Y-5L | Baseline, Week 26
Change in Homeostasis Model Assessment of Beta Cell Function (HOMA-B) | Baseline, Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (46):
- United States (39):
  - University of Arizona, Tucson, Arizona
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Division of Endocrinology, Diabetes, and Metabolism, Los Angeles, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital of Colorado, Denver, Colorado
  - Yale Diabetes Research, New Haven, Connecticut
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Nemours Children's Health, Jacksonville, Florida
  - D&H National Research Centers, Inc, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - D&H Tamarac Research Center, LLC, Tamarac, Florida
  - University of South Florida, Tampa, Florida
  - Children's Healthcare of Atlanta - Center for Advanced Pediatrics, Atlanta, Georgia
  - Centricity Research Columbus Endocrinology, Columbus, Georgia
  - St. Luke's Children's Endocrinology and Diabetes, Boise, Idaho
  - University of Illinois at Chicago, Chicago, Illinois
  - Center for Diabetes and Metabolic Diseases Indiana University, Indianapolis, Indiana
  - University of Iowa Stead Family Children's Hospitals, Iowa City, Iowa
  - Norton Children's Endocrinology, Louisville, Kentucky
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - WBMD Pediatrics, Buffalo, New York
  - Cohen Children's Medical Center Division of Pediatric Endocrinology, Hyde Park, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - UNC Children's Hospital, Chapel Hill, North Carolina
  - Childrens Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Childrens Outpatient Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St Christophers Hospital For Children, Philadelphia, Pennsylvania
  - Prisma Health Pediatric Endocrinology, Columbia, South Carolina
  - Research Institute of Dallas, Dallas, Texas
  - Texas Childrens Hospital, Houston, Texas
  - UT Health Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Wisconsin - Milwaukee Campus, Milwaukee, Wisconsin
- Argentina (5):
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - INECO Neurociencias Oroño, Rosario
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán
  - Go Centro Medico San Nicolás, San Nicolás
- Mexico (2):
  - Hospital Angeles (HA) - Puebla, Puebla City
  - Arké SMO S.A de C.V, Veracruz

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Dulaglutide (LY2189265) 3.0 mg and 4.5 mg in Pediatric Participants with Type 2 Diabetes Mellitus (AWARD-PEDS PLUS) — https://trials.lilly.com/en-US/trial/561355